CLINICAL TRIAL: NCT05890872
Title: A Clinical Study of Aliya™ Pulsed Electric Fields (PEF) Delivered Prior to Standard of Care Treatment for Advanced Cancer
Brief Title: Aliya™ Pulsed Electric Fields (PEF) for Advanced Cancer
Acronym: AFFINITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galvanize Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-00018
Record Dates: First submitted 2023-05-05; First posted 2023-06-06 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Lung Neoplasm Malignant
Keywords: Lung Neoplasms; Thoracic Neoplasms; Immunologic Factors
MeSH Terms: conditions — Lung Neoplasms; Thoracic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Aliya PEF (Experimental): Pulsed electric field treatment using the Aliya System
  Interventions: Device: Aliya Pulsed Electric Fields (PEF)

INTERVENTIONS:
Device: Aliya Pulsed Electric Fields (PEF) — Percutaneous or Endobronchial PEF

SUMMARY:
The goal of this clinical trial is to evaluate safety of delivering Aliya PEF in patients with metastatic cancer within the lungs or stage IV non-small cell lung cancer (NSCLC) who are treatment-naïve and indicated for first-line standard of care (SOC) cancer therapy.

DETAILED DESCRIPTION:
The Aliya Treatment System is designed to deliver therapeutic PEF energy to target tissues, via either a percutaneous or bronchoscopic approach. In order to evaluate the therapeutic potential of PEF delivered via the Aliya Treatment System as an interventional treatment, this clinical trial will evaluate the safety of delivering Aliya PEF in non-surgical advanced stage disease treatment-naïve patients indicated for diagnostic biopsy and first line (1L) standard of care (SOC) therapy. Additionally, this study will examine the safety of adding PEF treatment to the care pathway for patients with metastatic cancer to the lung or stage IV NSCLC and further assess the potential immune modulation and treatment effect of PEF for providing benefit to oncological patients, as outlined below.

ELIGIBILITY:
Inclusion Criteria:

* Patient has suspected or confirmed metastatic cancer within the lungs, or stage IV non-small cell lung cancer (NSCLC) requiring biopsy.
* Patient has radiologically documented suspected, or confirmed tumor(s) that are ≤ 5 cm in longest diameter and deemed by the investigator to be suitable per study procedural guidelines for treatment with PEF.
* Patient is deemed eligible to receive 1L SOC therapy for their malignancy.
* In the opinion of the investigator, the patient is not a surgical candidate for curative intent, or the patient has refused surgery.
* Life expectancy ≥ 6 months.

Exclusion Criteria:

* Patient has received any prior cancer therapy for current tumor(s) to be treated with PEF.
* Patient is scheduled to receive investigational therapies (including device-based therapy) that may interfere with the study endpoints while on this study.
* Patient has clinical evidence of leptomeningeal disease or brain metastases that require SOC treatment within 4 weeks post-PEF treatment.
* Patient with active, known, or suspected autoimmune disease.
* Patient with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Patient has received systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 30 days prior to study enrollment. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease.
* Patient has any history of primary immunodeficiency.
* Patient has clinical signs or symptoms of active tuberculosis infection.
* Patient has documented evidence of acute hepatitis or has an active or uncontrolled infection.
* Patient has undergone major surgery (excluding placement of vascular access) within 28 days prior to study enrollment or has planned major surgeries while enrolled in the study,

Other protocol defined inclusion/exclusion criteria apply

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Device and Procedure related serious adverse events | 30 days post PEF
  The rate of study device-related and/or PEF procedure-related serious adverse events (SAEs)
Percentage of subjects whose SOC cancer treatment was not cancelled or postponed | 1 year Post PEF
  The percentage of subjects whose SOC cancer treatment was not cancelled or postponed due to a PEF device- or procedure-related AE

SECONDARY OUTCOMES:
Procedural success | Day of procedure
  The frequency with which physicians can deliver PEF energy to intended targets
Anesthesia Type Usage | During PEF procedure
  Anesthesia Type Usage
PEF Target Location | During PEF procedure
  Anatomic lung region treated with PEF
Initiation of first-line (1L) SOC therapy following PEF treatment | 12 months
  Time to initiate first-line (1L) SOC therapy following PEF treatment

CONTACTS AND LOCATIONS:
Overall Officials: William Krimsky, MD, Study Chair — Chief Medical Officer
Locations (5):
- United States (5):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Weill Cornell Medicine | New York-Presbyterian, New York, New York
  - FirstHealth of the Carolinas, Inc., Pinehurst, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No